CLINICAL TRIAL: NCT07368998
Title: A Phase II, Randomized, Open-Label Study Evaluating Two Inavolisib Dose Levels in Combination With Fulvestrant in Participants With PIK3CA-Mutated, HR-Positive, HER2-Negative Locally Advanced or Metastatic Breast Cancer
Brief Title: To Study the Effect of Inavolisib in Combination With Fulvestrant in Participants With Breast Cancer
Acronym: optINAVO
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WO46063; 2025-522805-39-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-22; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — inavolisib; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Inavolisib Dose A plus Fulvestrant (Experimental): Participants will recieve an inavolisib tablet orally (PO) along with fulvestrant as an intramuscular (IM) injection.
  Interventions: Drug: Inavolisib; Drug: Fulvestrant
- Inavolisib Dose B plus Fulvestrant (Experimental): Participants will recieve an inavolisib tablet PO along with fulvestrant as an IM injection.
  Interventions: Drug: Inavolisib; Drug: Fulvestrant

INTERVENTIONS:
Drug: Inavolisib — Participants will receive Inavolisib as per the schedule given in the protocol.
Drug: Fulvestrant — Participants will receive Fulvestrant as per the schedule given in the protocol.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of inavolisib in combination with fulvestrant compared with inavolisib in combination with fulvestrant in participants with PIK3CA-mutated, HR-positive, HER2-negative locally advanced or metastatic breast cancer (LA/mBC) in the post-cyclin-dependent kinase inhibitor (CDKi) setting.

ELIGIBILITY:
Inclusion Criteria:

* Documented ER +/ HER2- tumor according to American Society of Clinical Oncology/College of American Pathologists (ASCO/CAP) guidelines
* Disease progression after or during treatment with a combination of CDK4/6i and endocrine therapy: <= 1 prior lines of systemic therapy in the locally advanced (recurrent or progressed) or metastatic setting
* Measurable or evaluable disease per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1)
* Participants for whom endocrine-based therapy is recommended and treatment with cytotoxic chemotherapy is not indicated at time of entry into the study, as per national or local treatment guidelines
* Confirmation of biomarker eligibility: presence of >= 1 study-eligible PIK3CA mutation
* Life expectancy of > 6 months
* Ability, in the investigator's judgment, and willingness to comply with all study -related procedures, including completion of patient-reported outcomes

Exclusion Criteria:

* Metaplastic breast cancer
* Prior treatment with chemotherapy in the recurrent locally advanced/metastatic setting
* Type 2 diabetes requiring ongoing systemic treatment at the time of study entry; or any history of Type 1 diabetes
* Prior treatment with PI3K/Akt/mTOR inhibitors in the recurrent locally advanced/metastatic setting
* Requirement for daily supplemental oxygen
* Symptomatic active lung disease, including pneumonitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-02-27 (Estimated); Primary Completion 2028-10-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Objective Response Rate (ORR) | Up to approximately 2 years
Percentage of Participants With Treatment Emergent Adverse Events (TEAEs) | Up to approximately 2 years

SECONDARY OUTCOMES:
Duration of Response (DOR) | Up to approximately 2 years
Time to Response (TTR) | Up to approximately 2 years
Progression-free Survival (PFS) | Up to approximately 2 years
Percentage of Participants With Treatment Discontinuation due to Adverse Events | Up to approximately 2 years
Number of Participants Reporting Presence, Frequency, Severity and/or Degree of Interference With Daily Activities of Symptomatic Treatment Toxicities as Assessed by NCI Patient-Reported Outcomes Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Up to approximately 2 years
Percentage of Participants Reporting Presence and Frequency of Selected Hyperglycemia Symptoms as Assessed by European Organisation for Research and Treatment of Cancer (EORTC) IL382 | Up to approximately 2 years
Percentage of Participants Reporting Each Response Option at Each Time Point for the Treatment Side-Effect Bother Item General Population, Question 5 (GP5) From the Functional Assessment of Cancer Therapy - General (FACT-G) Questionnaire | Up to approximately 2 years
Change from Baseline in Symptomatic Treatment-Related Toxicities as Assessed Through use of the PRO-CTCAE | Baseline, Up to approximately 2 years
Change from Baseline in Selected Hyperglycemia Symptoms as Assessed by EORTC IL382 | Baseline, Up to approximately 2 years
Change from Baseline in Treatment Side-effect Bother as Assessed Through use of the FACT-G GP5 Item | Baseline, Up to approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing